CLINICAL TRIAL: NCT04231266
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy of ManNAc in Subjects With GNE Myopathy
Brief Title: Multi-Center Study of ManNAc for GNE Myopathy
Acronym: MAGiNE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leadiant Biosciences, Inc. (Industry)
Collaborators: Brigham and Women's Hospital (Other); National Human Genome Research Institute (NHGRI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); NIH (NIAMS and NIND) as part of NeuroNext (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN109; 1U01AR070498-01A1 (NIH)
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: GNE Myopathy
Keywords: GNE Myopathy; Hereditary Inclusion Body Myopathy (HIBM); Distal Myopathy with Rimmed Vacuoles (DMRV); Nonaka Myopathy; Inclusion Body Myopathy type 2 (IBM-2)
MeSH Terms: conditions — Distal myopathy, Nonaka type | interventions — N-acetylmannosamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ManNAc (Active Comparator): Oral ManNAc will be administered at a dose of 4 grams three times daily (total of 12 grams daily).
  Interventions: Drug: ManNAc
- Placebo (Placebo Comparator): Oral Placebo will be administered three times daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ManNAc — Oral N-acetyl-D-mannosamine monohydrate (ManNAc)
  Other Names: N-acetyl-D-mannosamine monohydrate
  Arms: ManNAc
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
GNE myopathy is a rare genetic muscle disease characterized by progressive muscle atrophy and weakness. The disease is caused by mutations in the gene that encodes the enzyme that initiates and regulates N-acetylneuraminic acid (Neu5Ac) biosynthesis and glycan sialylation. Currently, there is no therapy available for this disease. N-Acetylmannosamine (ManNAc), an orphan drug in development for GNE myopathy, is an uncharged monosaccharide and the first committed precursor in Neu5Ac biosynthesis. In this randomized, double-blind, placebo-controlled trial the efficacy and long-term safety of ManNAc will be evaluated in subjects with GNE myopathy.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, multi-center study to evaluate the long-term safety and clinical efficacy of ManNAc in subjects with GNE myopathy.

A total of 51 eligible subjects will be randomized in a 2:1 ratio to receive either ManNAc at 4 g three times daily (total of 12 g/day) or placebo. Subjects will have follow-up visits every 6 months (±7 days) and take study drug for a minimum of 24 months, until their final study visit . The final on-site study visit for a subject is the last expected 6-month follow-up visit that occurs prior to the time the last randomized subject is expected to reach 24 months (extended follow-up).

Subjects will undergo screening and baseline evaluations that include clinical laboratory tests, Quantitative Muscle Assessment (QMA), the Inclusion Body Functional Myositis Rating Scale (IBMFRS), and other patient-reported outcomes (PROs), and rehabilitation medicine functional assessments. Follow-up evaluations will occur every six months following baseline, until 24 months after randomization of the last subject. Phone follow-up will occur every month without a clinic visit for the duration of the trial, and the last visit for each subject will be followed by phone follow-up 1 month after the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject should be 18-70 years of age at the time of enrollment, inclusive, and of either gender.
2. Subject has a diagnosis of GNE myopathy based upon a consistent clinical course and biallelic GNE gene mutations that classify as pathogenic or likely pathogenic according to American College of Medical Genetics and Genomics (ACMG) guidelines.
3. Subjects must have 10.00-65.99% of predicted muscle strength measured by QMA at screening in at least one of the selected muscle groups (ankle dorsiflexion, knee flexion, grip, shoulder abduction and elbow flexion).
4. Subject has the ability to travel to the Clinical Trial Site for visits.
5. Subjects must be able to communicate effectively with study staff and understand the requirements of the protocol without translators.
6. Subject must be able to comply with requirements of the protocol, including blood collection, drug administration, and muscle strength assessments.
7. Women of childbearing potential must be willing to use an effective method of contraception for the duration of the trial. It is recommended that male subjects follow birth control measures for the duration of the trial.
8. Subject must be able to provide informed consent.

Exclusion Criteria:

1. Subject had an infection or medical illness requiring intravenous antibiotics or hospitalization within 30 days prior to the baseline/randomization visit.
2. Subject has another comorbid condition which may affect physical function.
3. Subject has a psychiatric illness or neurological disease that would interfere with the ability to comply with the requirements of this protocol.
4. Subject with hepatic laboratory parameters (AST, ALT, GGTP), equal to or greater than 3 times the upper limit of normal at screening.
5. Subject with existing renal dysfunction, as defined by glomerular filtration rate (GFR) less than 60 mL/min/1.73 m2 at screening.
6. Subject is anemic (defined as Hematocrit <30%) or has platelets <75 x 10^3/µL or white blood cell count less than 3 x 10^3/µL at screening.
7. Subject shows evidence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, metabolic, or gastrointestinal disease, or has a condition that requires immediate surgical intervention.
8. Subject is pregnant or breastfeeding at any time during the study.
9. Subject has received treatment with another investigational drug, investigational device, or approved therapy for investigational use less than 90 days prior to screening.
10. Subject has received any dose of ManNAc, sialic acid, intravenous immunoglobulin (IVIG), and/or other compounds containing, or that can be metabolized into sialic acid, within 6 months prior to enrollment as reported by subject at the time of screening.
11. Subject has received stem cell therapy or gene therapy within 1 year prior to screening.
12. Subject has hypersensitivity to ManNAc or erythritol or in the judgment of the investigator, has a condition that places the subject at increased risk for adverse effects.
13. The presence of persistent diarrhea or malabsorption that could interfere with the subject's ability to absorb drugs or to tolerate ManNAc therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-06-27 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Muscle strength of ankle dorsiflexion, knee flexion, knee extension, shoulder abduction, elbow flexion and grip measured by fixed-frame Quantitative Muscle Assessment (QMA) | Minimum 2 years, until 24 months from randomization of last subject
  The primary endpoint is the change in muscle strength decline under treatment compared to placebo. The primary analysis is based on the disease progression ratio (γ) comparing the rate of progression from baseline until last visit, under placebo to that under treatment.

SECONDARY OUTCOMES:
Inclusion Body Myositis Functional Rating Scale (IBMFRS) | Minimum 2 years, until 24 months from randomization of last subject
  Change in patient-reported function as measured by the Inclusion Body Myositis Functional Rating Scale (IBMFRS).

OTHER OUTCOMES:
Adverse Events | Minimum 2 years, until 24 months from randomization of last subject
  Safety and tolerability will be evaluated by comparing the frequency of adverse events (AEs) across groups, collected using information from in-person assessments, clinical laboratory tests, vital signs, electronic diary reports, and physical examinations.
Correlation muscle strength measured Exploratory GNEM Functional Questions (ExGNEM) | Minimum 2 years, until 24 months from randomization of last subject
  Evaluate the effect of ManNAc on patient-reported physical functioning assessed by ExGNEM, a six-question rating scale that assesses lower body function.
Adult Myopathy Assessment Tool | Minimum 2 years, until 24 months from randomization of last subject
  Evaluate the effect of ManNAc on physical function as measured by the Adult Myopathy Assessment Tool (AMAT), a 13-item standardized test that assesses physical performance, to be performed at baseline and every 6 months thereafter until completion of the study.
Six-Minute Walk Test | Minimum 2 years, until 24 months from randomization of last subject
  Evaluate the effect of ManNAc on physical function as measured by the Six-Minute Walk Test (whenever possible) to be performed at baseline and every 6 months thereafter until completion of the study.
Timed Up and Go Test | Minimum 2 years, until 24 months from randomization of last subject
  Evaluate the effect of ManNAc on physical function as measured by the Timed Up and Go, performance test to evaluate functional mobility, to be performed at baseline and every 6 months thereafter until completion of the study.
Functional Reach Test | Minimum 2 years, until 24 months from randomization of last subject
  Evaluate the effect of ManNAc on physical function as measured by the Functional Reach, a measure of stability, to be performed at baseline and every 6 months thereafter until completion of the study.
Jebsen Hand Function Test | Baseline and every 12 months thereafter
  Evaluate the effect of ManNAc on physical function as measured by the Jebsen Hand Function Test, a performance measure which assesses unilateral hand function, to be performed at baseline and every 6 months thereafter until completion of the study.
Inclusion Body Myositis Functional Rating Scale | Minimum 2 years, until 24 months from randomization of last subject
  Evaluate effect of ManNAc on activities of daily living (ADLs) compared to placebo as measured by the Inclusion Body Myositis Functional Rating Scale (IBMFRS), a patient-reported outcome completed at baseline, and every 6 months thereafter until completion of the study.
Human Activity Profile | Minimum 2 years, until 24 months from randomization of last subject
  Evaluate effect of ManNAc on activities of daily living (ADLs) compared to placebo as measured by the Human Activity Profile, a patient-reported outcome completed at baseline, and every 6 months thereafter until completion of the study.
Activities-specific Balance Confidence (ABC) scale | Minimum 2 years, until 24 months from randomization of last subject
  Evaluate effect of ManNAc on activities of daily living (ADLs) compared to placebo as measured by the Activities-specific Balance Confidence (ABC) scale, a patient-reported outcome completed at baseline, and every 6 months thereafter until completion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A. Amato, MD, Principal Investigator — Brigham and Women's Hospital; Francis Rossignol, MD, Principal Investigator — National Institutes of Health (NIH)
Locations (10):
- United States (10):
  - UCLA, Los Angeles, California
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Medical Center, Kansas City, Kansas
  - NIH Clinical Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Ohio State University, Wexner Medical Center, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quintana M, Shrader J, Slota C, Joe G, McKew JC, Fitzgerald M, Gahl WA, Berry S, Carrillo N. Bayesian model of disease progression in GNE myopathy. Stat Med. 2019 Apr 15;38(8):1459-1474. doi: 10.1002/sim.8050. Epub 2018 Dec 3. PMID 30511500
- [Background] Carrillo N, Malicdan MC, Huizing M. GNE Myopathy: Etiology, Diagnosis, and Therapeutic Challenges. Neurotherapeutics. 2018 Oct;15(4):900-914. doi: 10.1007/s13311-018-0671-y. PMID 30338442
- [Background] Xu X, Wang AQ, Latham LL, Celeste F, Ciccone C, Malicdan MC, Goldspiel B, Terse P, Cradock J, Yang N, Yorke S, McKew JC, Gahl WA, Huizing M, Carrillo N. Safety, pharmacokinetics and sialic acid production after oral administration of N-acetylmannosamine (ManNAc) to subjects with GNE myopathy. Mol Genet Metab. 2017 Sep;122(1-2):126-134. doi: 10.1016/j.ymgme.2017.04.010. Epub 2017 Apr 26. PMID 28641925
- See also: Study NN109/MAGiNE website — https://neuronext.org/projects/nn109-magine